CLINICAL TRIAL: NCT00686244
Title: Effect of Personal and IT Based Training to Performance, Metabolic Profil and Quality of Life by Patients With Metabolic Syndrome
Brief Title: IT-Based Training in Metabolic Syndrome
Acronym: SPRINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Martin Halle, Ph.D., Department of Sports Medicine, Klinikum rechts der Isar, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FKZ01FD0609
Record Dates: First submitted 2008-05-21; First posted 2008-05-29 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; physical activity; overweight; malnutrition; prevention
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity; Overweight; Malnutrition | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training Group (Experimental): Combined 3-monthly endurance- (3x/week) and strength training (2x/week) with moderate beginning and continuous increase of volume, duration and intensity, orientated on metabolic equivalents (MET).
  Main sport: walking, walk and cycling. Addition with other activities are possible up to once a week to achieve the basal metabolism
  Interventions: Other: Combined 3-monthly endurance and strength training
- Control Group (No Intervention): No guided training. Exercise optional after detailed consulting and handing over an information dossier for adequate physical activity.

INTERVENTIONS:
Other: Combined 3-monthly endurance and strength training — Combined 3-monthly endurance- (3x/week) and strength training (2x/week) with moderate beginning and continuous increase of volume, duration and intensity, orientated on metabolic equivalents (MET).
  Main sport: walking, walk and cycling. Addition with other activities are possible up to once a week to achieve the basal metabolism
  Arms: Training Group

SUMMARY:
Prospective, randomized, single center, controlled intervention study to investigate the effect of a systematic combined personal and IT-based training on the outcome of patients with metabolic syndrome.

DETAILED DESCRIPTION:
The study settles in the field of primary prevention and aims to change lifestyle of patients with metabolic syndrome with a new combination of personal and IT-based training specially designed für obese people with risk factors. Procedures that are similar for all participants are summarized in a training program whereas individual aspects of physical activity like initial education and exercise tests are still performed by doctors and trainers. Before and after three months of training anthropometric parameters, laboratory and exercise capacity are examined and analyzed. The intervention group is characterized by a predetermined exercise program whereas the control group is allowed to practise without detailed instructions. The practicability and the effect on health status of the combined personal and IT-based training in the intervention group is compared with the independent training of the control group. After 6 months and again after 12 months the measurements are repeated to evaluate a lasting effect of the program.

ELIGIBILITY:
Inclusion Criteria:

* males and females between 20 and 60 years
* Staff of the Fa. BMW
* written informed consent after detailed education
* BMI 25-35 kg/m2
* ≤ 1x/week sport respectively exercise
* metabolic syndrome (at least 3 of 5 criteria)

Exclusion Criteria:

* > 1x/week physical activity
* BMI < 25 kg/m2 or > 35 kg/m2
* Florid acute or chronic disease of any kind prohibiting regular physical activity
* Diabetes mellitus
* pregnancy or lactation
* Drug or alcohol abuse

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of a combined personal and IT- based training on the performance at the metabolic anaerobe barrier of patients with impending or manifest metabolic syndrome compared to a control group with conventional consulting | 12 months

SECONDARY OUTCOMES:
Evaluation of the effect of IT based training on metabolic parameters | 12 months
Evaluation of the efficacy of IT based training to an increase of activity by patients with impending or manifest metabolic syndrome | 12 months
Change in quality of life and subjective assumption of health sensation | 12 months
Change in anthropometric parameters | 12 months
Raise of maximum performance (max. ergometric performance) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, P.D., Principal Investigator — Department of Sports Medicine, Klinikum rechts der Isar, Technical University of Munich
Locations (1):
- Lehrstuhl für Praeventive und Rehabilitative Sportmedizin Klinikum Rechts der Isar, Technical University of Munich, Munich, Germany

REFERENCES:
- [Background] Ainsworth BE, Anderson LA, Becker DM, Blalock SJ, Brown DR, Brownson RC, Brownstein N, Cornell CE, Devellis BM, Finnegan LP, Folger S, Fulton JE, Groff JY, Herman C, Jones D, Keyserling TC, Matson Koffman D, Lewis C, Masse LC, McKeown RE, Orenstein D, Spadaro AJ; Women's Health Initiative Community Prevention Study Collaborators. Observations from the CDC. Community Prevention Study: contributions to women's health and prevention research. J Womens Health Gend Based Med. 2001 Dec;10(10):913-20. doi: 10.1089/152460901317193495. No abstract available. PMID 11788102
- [Background] Bullinger M, Kirchberger I. SF-36. Fragebogen zum Gesundheitszustand. Göttingen, Hogrefe 1998
- [Background] Centers for disease control. Overweight and obesity. www.cdc.gov/nccdphp/dnpa/obesity/trend/maps/index.htm
- [Background] Chisholm DM, Collis ML, Kulak LL, Davenport W, Gruber N. Physical activity readiness. Br Col Med J 17(1975);375-78
- [Background] Deutsches Netzwerk für Betriebliche Gesundheitsförderung. www.dnbgf.de
- [Background] Frey I, Berg A, Grathwohl D, Keul J. [Freiburg Questionnaire of physical activity--development, evaluation and application]. Soz Praventivmed. 1999;44(2):55-64. doi: 10.1007/BF01667127. German. PMID 10407953
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Konig D, Bonner G, Berg A. [The role of adiposity and inactivity in primary prevention of cardiovascular disease]. Herz. 2007 Oct;32(7):553-9. doi: 10.1007/s00059-007-3019-7. German. PMID 17972028
- [Background] Nationale Verzehrstudie II. Bundesministerium für Ernährung, Landwirtschaft, und Verbraucherschutz. www.was-esse-ich.de
- [Background] Parizkova J, Buzkova P. Relationship between skinfold thickness measured by Harpenden caliper and densitometric analysis of total body fat in men. Hum Biol. 1971 Feb;43(1):16-21. No abstract available. PMID 5556752
- [Background] Statistisches Bundesamt. www.destatis.de
- [Background] Sullivan PW, Morrato EH, Ghushchyan V, Wyatt HR, Hill JO. Obesity, inactivity, and the prevalence of diabetes and diabetes-related cardiovascular comorbidities in the U.S., 2000-2002. Diabetes Care. 2005 Jul;28(7):1599-603. doi: 10.2337/diacare.28.7.1599. PMID 15983307
- [Background] Vatten LJ, Nilsen TI, Romundstad PR, Droyvold WB, Holmen J. Adiposity and physical activity as predictors of cardiovascular mortality. Eur J Cardiovasc Prev Rehabil. 2006 Dec;13(6):909-15. doi: 10.1097/01.hjr.0000239463.80390.52. PMID 17143122
- [Background] Graham I, Atar D, Borch-Johnsen K, Boysen G, Burell G, Cifkova R, Dallongeville J, De Backer G, Ebrahim S, Gjelsvik B, Herrmann-Lingen C, Hoes A, Humphries S, Knapton M, Perk J, Priori SG, Pyorala K, Reiner Z, Ruilope L, Sans-Menendez S, Op Reimer WS, Weissberg P, Wood D, Yarnell J, Zamorano JL, Walma E, Fitzgerald T, Cooney MT, Dudina A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Funck-Brentano C, Filippatos G, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Altiner A, Bonora E, Durrington PN, Fagard R, Giampaoli S, Hemingway H, Hakansson J, Kjeldsen SE, Larsen ML, Mancia G, Manolis AJ, Orth-Gomer K, Pedersen T, Rayner M, Ryden L, Sammut M, Schneiderman N, Stalenhoef AF, Tokgozoglu L, Wiklund O, Zampelas A; European Society of Cardiology (ESC); European Association for Cardiovascular Prevention and Rehabilitation (EACPR); Council on Cardiovascular Nursing; European Association for Study of Diabetes (EASD); International Diabetes Federation Europe (IDF-Europe); European Stroke Initiative (EUSI); International Society of Behavioural Medicine (ISBM); European Society of Hypertension (ESH); European Society of General Practice/Family Medicine (ESGP/FM/WONCA); European Heart Network (EHN). European guidelines on cardiovascular disease prevention in clinical practice: executive summary. Fourth Joint Task Force of the European Society of Cardiology and other societies on cardiovascular disease prevention in clinical practice (constituted by representatives of nine societies and by invited experts). Eur J Cardiovasc Prev Rehabil. 2007 Sep;14 Suppl 2:E1-40. doi: 10.1097/01.hjr.0000277984.31558.c4. No abstract available. PMID 17726406